CLINICAL TRIAL: NCT02082327
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of Migalastat Hydrochloride Given Intravenously to Healthy Volunteers With an Open-Label, Randomized, Two-Way Crossover Arm
Brief Title: A Phase 1 Study To Evaluate the Safety of Migalastat Hydrochloride Given Intravenously to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT1001-018; 2013-005553-75 (EudraCT Number)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-04

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Fabry; Lysosomal storage disorders; LSD; Amicus; migalastat HCl; migalastat; AT1001
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases | interventions — migalastat; larazotide acetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.3 mg/kg (Experimental): IV infusion of migalastat HCl or placebo
  Interventions: Drug: IV migalastat HCl; Drug: IV placebo
- 1 mg/kg (Experimental): IV infusion of migalastat HCl or placebo
  Interventions: Drug: IV migalastat HCl; Drug: IV placebo
- 10 mg/kg (Experimental): IV infusion of migalastat HCl or placebo
  Interventions: Drug: IV migalastat HCl; Drug: IV placebo
- 150 mg IV (Experimental): 150 mg single IV infusion
  Interventions: Drug: IV migalastat HCl; Drug: oral migalastat HCl
- 150 mg oral (Experimental): 150 mg single oral dose
  Interventions: Drug: IV migalastat HCl; Drug: oral migalastat HCl

INTERVENTIONS:
Drug: IV migalastat HCl
  Other Names: AT1001
Drug: IV placebo
  Other Names: Sodium Chloride 0.9%
  Arms: 0.3 mg/kg; 1 mg/kg; 10 mg/kg
Drug: oral migalastat HCl
  Other Names: AT1001
  Arms: 150 mg IV; 150 mg oral

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of IV migalastat HCl alone and to determine absolute bioavailability for oral migalastat HCl as compared to IV administered migalastat HCl in healthy volunteers. The data from this study will help us understand how migalastat works in the body and will help us determine what would be an effective dose in future studies with migalastat hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 45 years of age.
* Body weight range ≥ 50 kg ≤ 100 kg and BMI within the range 18.5 - 29.9 kg/m2.
* Healthy as determined by a responsible and experienced physician, based on a medial evaluation.
* Male and female subjects of childbearing potential agree to adhere to the contraception requirements.
* Capable of giving written informed consent.

Exclusion Criteria:

* History of sensitivity to migalastat HCl or related iminosugars (eg, miglitol, miglustat), or other significant drug allergy.
* Past medical history, or physical examination findings, of clinically significant abnormalities that may put the subject at risk or interfere with outcome variables.
* Positive pre-study drug/alcohol screen.
* Pregnant or lactating females.
* The subject has participated in a clinical trial and has received an investigational product within 60 days prior to the first dosing day in the current study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics of migalastat | Pre-dose, 0.25, 0.5, 1, 1.5, 2.0, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48
  To investigate the effect on the body of migalastat following a single 2 hour IV infusion in healthy subjects.
Safety and tolerability of migalastat | 48 hours
  Adverse events, clinical laboratory test values, vital signs, ECG, physical examinations

SECONDARY OUTCOMES:
Plasma pharmacokinetics of migalastat | Pre-dose, 0.25, 0.5, 1, 1.5, 2.0, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48
  To assess the dose proportionality of migalastat following a single 2 hour IV infusion
Urinary pharmacokinetics | Pre dose, between 0-6, 6-12 and 12-24 hours after start of infusion
  To estimate the urinary excretion of unchanged migalastat following a single 2 hour IV infusion in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Research, Study Director — Amicus Therapeutics
Locations (1):
- PRA International, Groningen, Netherlands